CLINICAL TRIAL: NCT02104128
Title: Effects of Bupropion in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Bup_dep_1; 13/SC/0569 (Other: NRES Ethics Committee); OxH 1005 (Other: Oxford Health R&D)
Record Dates: First submitted 2014-03-24; First posted 2014-04-04 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Depression
Keywords: Anhedonia; Dopamine; Bupropion; fMRI; emotional processing; reward
MeSH Terms: conditions — Depression; Anhedonia | interventions — Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depressed patient given bupropion (Experimental): All depressed patients will be given open label bupropion
  Interventions: Drug: Bupropion
- Control pts given no intervention (No Intervention): Control participants will be assessed at the same time points as the depressed group, but will be given no drug

INTERVENTIONS:
Drug: Bupropion — Bupropion MR will be given open label to all participants in the depression group. Participants will receive 150mg od for one week. The dose will then be increased to 150mg bd for the following 5 weeks. Participants in the control group will recieve no drug. Note that the study is not assessing the safety or efficacy of buprion-- it is using bupropion to assess the neural effects of altering central dopaminergic function in depressed patients.
  Other Names: Zyban
  Arms: Depressed patient given bupropion

SUMMARY:
This study will investigate the role of dopaminergic neural systems in the symptoms and treatment of depression. 40 patients who meet DSM-IV criteria for a diagnosis of depression will be compared to a matched sample of healthy controls. The depressed group will receive open label treatment with Bupropion MR (150mg bd) for 6 weeks. The control group will receive no treatment. All participants will be assessed before treatment, after 2 weeks treatment and at 6 weeks treatment. The outcomes assessed will be 1) fMRI estimates of neural response to reward to emotionally valenced stimuli (1st and 2nd assessments), 2) computer based measures of emotional processing (all assessments) and 3) standardised questionnaire measures of depressive symptoms (all assessments). The primary study hypothesis is that altering central dopamine using Bupropion will lead to altered neural responses to rewarding stimuli in the depressed patients (i.e. comparing fMRI outcomes between assessment visits 1 and 2). A secondary hypothesis is that this neural change will predict subsequent symptom response to the bupropion (i.e. comparing symptom scores between assessment visits 1 and 3), Lastly, the study will test the hypothesis that baseline differences in reward circuitry will be particularly associated with symptoms of anhedonia (the inability to experience pleasure).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have signed an informed consent document indicating they understand the purpose of the study and the procedures required for the study and are willing to participate by complying with the study procedures and restrictions
* Participants will be male or female and aged between 18 and 50
* Participants will have a Body Mass Index (BMI) 18 to 36 kg/m2 (inclusive) at the Screening Visit.
* The MDD participants must satisfy a diagnosis of MDD as determined by structured clinical interview for DSM-V (SCID) conducted by a psychiatrist. The MDD subtypes characterized under DSM-V also will be determined for use during post hoc tests aimed at characterizing further the heterogeneity extant within the MDD population.
* Participants must be sufficiently fluent in English to complete the emotional and reward tasks.

Exclusion Criteria:

* Current use of psychotropic medication or electroconvulsive therapy (within three weeks of the baseline assessments) or psychological treatment (within 3 months of the baseline assessments)
* They are left handed (the site of brain activations vary depending on handedness)
* They are not fluent in English
* History of stimulant abuse (lifetime; e.g., amphetamine, cocaine), or of alcohol abuse within one year or of alcohol dependence within the lifetime.
* History of, or current medical conditions which in the opinion of the investigator may interfere with the scientific assessments or safety of the participant, including brain injury, epilepsy/seizures, severe hepatic cirrhosis and CNS tumour.
* Clinically significant abnormal values for liver function tests, clinical chemistry, urine drug screen, blood pressure measurement and ECG. It is expected that laboratory values will generally be within the normal range for the laboratory. NB clinical significance will be determined by a qualified study medic who will review the results and the participant.
* Current pregnancy or breastfeeding
* Smoker > 10 cigarettes per day or similar levels of tobacco consumption in other forms. History of smoking within 8 weeks of becoming abstinent.
* Any contraindication to MRI scanning, for example any metal implants in the body that include ferromagnetic objects in their bodies (e.g., metal implants, vessel clips, shrapnel injuries) or with implanted devices which may be damaged by the magnet (e.g., heart pacemakers).
* Participation in a psychological or medical study involving the use of medication within the last 3 months. Previous participation in any study involving the emotional test battery.
* Has clinically significant risk of suicidal behaviour.
* Medical conditions that may alter the hemodynamic parameters underlying the BOLD signal (e.g., inadequately treated hypertension, diabetes mellitus).

The following exclusion criteria apply specifically to the participants in the MDD group:

* Any known allergy, hypersensitivity or intolerance to bupropion or its excipients.
* Has any contraindication to the use of bupropion.
* Any medical contraindication, for example conditions or treatments that may alter the absorption of bupropion such as surgical treatments involving the gut.
* History of or current Axis 1 DSM-V psychiatric disorder (except depression or anxiety disorders such as specific phobia or social anxiety disorder for the MDD group and drug abuse subject to the criteria outlined below).The presence of co-morbid anxiety disorders will be recorded for potential use in post hoc exploratory analyses of the influence of such conditions on the outcome measures

The following criteria apply specifically to participants in the healthy control group:

• History of or current Axis 1 DSM-V psychiatric disorder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in haemodynamic (i.e. BOLD signal) response | Baseline and 2 weeks
  fMRI data collected during a reward and emotional coding task

SECONDARY OUTCOMES:
Change in questionnaire measures of subject mood and anhedonia | baseline, 2 and 6 weeks
  Standardised questionnaire measures of depressive symptoms and anhedonia.
Change in accuracy and reaction time | baseline, 2 and 6 weeks
  Behavioral responses during computer based tasks measures cognition

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Harmer, DPhil, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, Oxfordshire, United Kingdom